CLINICAL TRIAL: NCT07028398
Title: Nurse Follow-up to Reduce Inappropriate Emergency Department Utilization in Adult Patients Seen for Ambulatory Sensitive Conditions in CMSL Study 2
Brief Title: CMSL Ambulatory Sensitive Condition Nudge Study 2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Responsible Party: Principal Investigator, Amir Goren, Program Director, Geisinger Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2023-1716-2
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Behavioral Intervention; Emergency Department Visits; Nurse Care Coordination
Keywords: Nudge

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nurse Nudge (Experimental): Nurses in CMSL clinics will receive a notification to provide follow-up outreach (calls and/or patient portal messages) to patients after the patient receives an ambulatory sensitive diagnosis.
  Interventions: Behavioral: Nurse Nudge
- Control (No Intervention): Nurses in CMSL clinics will receive standard follow- up notifications, which may mean no notifications, after a patient has received an ambulatory sensitive diagnosis.

INTERVENTIONS:
Behavioral: Nurse Nudge — Nurses will be nudged to contact patients, which may increase the likelihood that the patient receives a post- appointment follow-up call and/or portal message.
  Arms: Nurse Nudge

SUMMARY:
The project aims to evaluate a nurse-led intervention to reduce inappropriate emergency department (ED) use among adult patients seen at Geisinger's Community Medicine Service Line (CMSL) clinics. The intervention occurs immediately following an appointment where a patient receives a diagnosis of an ambulatory sensitive condition (ASC; i.e., a condition considered to be a risk factor for near-term ED use). The evaluation will compare eligible patients with an ASC who were randomly assigned to receive follow-up outreach (patient portal message and/or call) from a nurse (who was automatically prompted via the Epic electronic health record system to initiate outreach) with those who were randomly assigned to receive standard care. Analyses will be intent-to-treat. The primary outcome is ED use in the week (i.e., 7 days) following the appointment.

We ran an earlier version of this intervention (NCT06798389). The current study is modified based on results and clinical guidance. Specifically, more conditions will be included as qualifying ASCs for enrollment. Patients under 30 will be excluded. And rather than calling all patients as in the original study, patient portal users may be contacted via the portal instead of or in addition to a phone call. Finally, in the first study, the intervention was differentially effective by age group (<45, 45-64, 65+). Our primary analysis will be conducted separately by age group, though we will also conduct an analysis combining across age groups.

We will run the study until we reach at least 4,330 patients in each of the following age groups: patients aged 30-45, patients aged 45-64, patients aged 65+. Therefore, our estimated sample size is at least 4,330x3 = 12,990.

We may be required to do an interim data pull and/or stop the study early at the direction of clinical or operational leaders.

ELIGIBILITY:
Inclusion Criteria:

* Age 30 years +
* Has a qualifying visit in CMSL with an ambulatory sensitive condition (ASC) encounter diagnosis

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12990 (Estimated)
Dates: Start 2025-05-29 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
ED Visit (yes/no) | within 7 days post-appointment
  Visited the ED (y/n)

OTHER OUTCOMES:
Nurse call to patient | Within 7 days post-appointment
  Nurse calls patient (y/n)
Nurse message to patient | Within 7 days post-appointment
  Nurse sends MyChart message to patient (y/n)
Nurse calls or sends message to patient | Within 7 days post-appointment
  Nurse calls or sends MyChart message to patient (y/n)

CONTACTS AND LOCATIONS:
Locations (1):
- Geisinger, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-11-18): https://cdn.clinicaltrials.gov/large-docs/98/NCT07028398/Prot_SAP_001.pdf